CLINICAL TRIAL: NCT01589146
Title: ONE WEEK VERSUS FOUR WEEK HEPARIN PROPHYLAXIS IN PATIENTS WITH COLORECTAL CANCER UNDERGOING LAPAROSCOPIC SURGERY: INCIDENCE OF VENOUS THROMBOEMBOLISM AND BLEEDING COMPLICATIONS. THE PRO-LAPS STUDY.
Brief Title: ONE WEEK VERSUS FOUR WEEK HEPARIN PROPHYLAXIS AFTER LAPAROSCOPIC SURGERY FOR COLORECTAL CANCER.
Acronym: PRO-LAPS I
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Cecilia Becattini, MD, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Unipg-CRU-01-2012
Record Dates: First submitted 2012-04-28; First posted 2012-05-01 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: The Primary Study Objective is to Assess the Efficacy and; Safety of Extended 4-week Heparin Prophylaxis Compared to; Prophylaxis Given for 8±2 Days After Planned Laparoscopic; Surgery for Colorectal Cancer.; The Clinical Benefit Will be Evaluated as the Difference in; the Incidence of VTE or VTE-related Death Occurring Within 30 Days; From Surgery in the Two Study Groups.
Keywords: colon-rectal cancer; heparin; prophylaxis; laparoscopy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- short heparin (No Intervention)
- extended heparin (Experimental)
  Interventions: Drug: Heparin, Low-Molecular-Weight

INTERVENTIONS:
Drug: Heparin, Low-Molecular-Weight — 4 weeks heparin prophylaxis
  Arms: extended heparin

SUMMARY:
Overall, only limited evidence exists regarding the clinical benefit of antithrombotic prophylaxis after laparoscopic surgery for cancer. Four studies reported on the incidence of venous thromboembolism (VTE) after laparoscopic surgery for cancer. These studies differ concerning study design, site of cancer, regimens for antithrombotic prophylaxis and reported incidence of VTE.

The aim of this multicenter, randomized study is to assess the clinical benefit of extended (4 weeks) compared to short (one week) heparin prophylaxis after laparoscopic surgery for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who had
* planned laparoscopic surgery for
* colorectal cancer will be included in the study provided no exclusion criteria will be found

Exclusion Criteria:

* age < 18 years
* surgery for non-cancer disease
* duration of surgery < 45 min
* other indication for anticoagulant therapy
* known cerebral metastases
* kidney or liver failure
* known hemorrhagic diathesis or high risk for bleeding
* history of intracerebral bleeding or neurosurgery within 6 months, history of heparin induced thrombocytopenia
* pregnancy or lactation
* refusal of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
symptomatic objectively confirmed VTE, asymptomatic ultrasonography-confirmed DVT or VTE-related death | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Internal and Cardiovascular Medicine - University of Perugia, Perugia, Italy

REFERENCES:
- [Derived] Vedovati MC, Becattini C, Rondelli F, Boncompagni M, Camporese G, Balzarotti R, Mariani E, Flamini O, Pucciarelli S, Donini A, Agnelli G. A randomized study on 1-week versus 4-week prophylaxis for venous thromboembolism after laparoscopic surgery for colorectal cancer. Ann Surg. 2014 Apr;259(4):665-9. doi: 10.1097/SLA.0000000000000340. PMID 24253138